CLINICAL TRIAL: NCT04593966
Title: Differences of Long-term Neurofunctional Outcomes in Pediatric and Adult Eloquent Region Cerebral Arteriovenous Malformation
Brief Title: Pediatric and Adult Cerebral Arteriovenous Malformation Neurofunctional Outcomes
Acronym: DOPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: yuanli Zhao (Other)
Collaborators: Peking University International Hospital (Other)
Responsible Party: Sponsor-Investigator, yuanli Zhao, Chairman of Neurosurgical center, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: KY 2019/0917
Record Dates: First submitted 2020-09-10; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Arteriovenous Malformation
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric AVM: 1. AVM patients' age under 18-years-old who underwent intervention in investigators' institution.
  2. Patients' lesions were located in eloquent and confirmed by image.
- Adult AVM: 1. AVM patients' age over 18-years-old who underwent intervention in investigators' institution.
  2. Patients' lesions were located in eloquent and confirmed by image.

SUMMARY:
Cerebral Arteriovenous malformations (AVMs) are abnormal tangles which are usually believed congenital. AVM can cause different symptoms depending on where it is located, but the most common symptoms are intracranial hemorrhage and seizure. Outcomes of AVM patients can be very different due to factors like the location of lesion, age, sex etc. Generally, more early the intervention was taken, the risk of adverse events would be lower. But the selection of surgical timing for pediatric AVM patients is hard to judge, due to children's cerebral vessels angioarchitecture can be still developing with their age. Some previous studies indicated that there is no difference in intervention outcomes between pediatric and adult AVM patients, so pediatric patients should undergo more aggressive intervention. DOPA study aims to compare the clinical intervention outcomes of both pediatric and adult patients with eloquent region cerebral arteriovenous malformations, helping to determine the treatment strategy.

DETAILED DESCRIPTION:
Follow-up: In the investigators' neurosurgical center, follow-up was conducted for all participants at the first 3-6 months and annually after discharge by clinical visit and telephone interview.

Study overview: DOPA will aim on outcomes of both pediatric and adult AVMs patients who underwent intervention in investigators' institution. Intervention strategies contains microsurgical resection, embolization, embolization + radiosurgery, and single-stage hybrid surgery (embolization + resection). Outcomes will be measured by a neurologist using Modified Rankin Scale (mRs). Participants' mRs<2 will be considered as a good outcome and investigators will keep follow-up with every patient for at least 3 years.

Sample size: About 300 patients will be enrolled in this study, and adults and children will account for half. All kinds of intervention will be included. The distribution of different strategies is excepted as: 30% resection, 20% embolization, 30% embolization + radiosurgery and 20% hybrid surgery.

Study endpoints: The patients' mRs, occlusion rate and complication will be evaluated at 2 weeks, discharge from hospital, 1 year and 3 years after the first-time intervention.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of AVM was confirmed with digital subtraction angiography (DSA) and/or magnetic resonance imaging(MRI).
* Patients had underwent interventions in our institution.
* AVMs were located in eloquent area.

Exclusion Criteria:

* Patients with multiple AVMs.
* Patients with hereditary hemorrhagic telangiectasia (HHT).
* Patients with missing clinical and imaging data.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with brain arteriovenous malformation which located in eloquent area.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-04-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
modified Ranking Scale score at 2 weeks after the operation | 2 weeks
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  No significant disability. Able to carry out all usual activities, despite some symptoms.
  Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Moderate disability. Requires some help, but able to walk unassisted. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Dead
modified Ranking Scale score when discharge | Discharge (assessed up to 10 days)
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  No significant disability. Able to carry out all usual activities, despite some symptoms.
  Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Moderate disability. Requires some help, but able to walk unassisted. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Dead
modified Ranking Scale score at 1 years after the operation | 1 years
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  No significant disability. Able to carry out all usual activities, despite some symptoms.
  Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Moderate disability. Requires some help, but able to walk unassisted. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Dead
modified Ranking Scale score at 3 years after the operation | 3 years
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  No significant disability. Able to carry out all usual activities, despite some symptoms.
  Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Moderate disability. Requires some help, but able to walk unassisted. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Dead

SECONDARY OUTCOMES:
Obliteration rate | At least 1 year, up to 3 years
  Confirmed by postoperative DSA or MRI/magnetic resonance angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Capital medical university affiliated Beijing Tiantan hospital, Beijing, Beijing Municipality, China